CLINICAL TRIAL: NCT00757692
Title: A Phase II Randomised Efficacy and Safety Study of Vandetanib (ZD 6474) in Combination With Bicalutamide Versus Bicalutamide Alone in Patients With Chemotherapy Naive Hormone Refractory Prostate Cancer.
Brief Title: Efficacy and Safety Study of Vandetanib (ZD 6474) in Combination With Bicalutamide Versus Bicalutamide Alone in Patients With Chemotherapy Naive Hormone Refractory Prostate Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OZM-011
Record Dates: First submitted 2008-09-19; First posted 2008-09-23 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Prostate Cancer
Keywords: Vandetanib (ZD6474); Hormone; Refractory; Prostate Cancer; Chemotherapy; Naïve
MeSH Terms: conditions — Prostatic Neoplasms | interventions — vandetanib; bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Vandetanib at 300 mg in combination with Bicalutamide at 50 mg will be administered orally, daily and continuously
  Interventions: Drug: Vandetanib
- B (Active Comparator): Bicalutamide at 50 mg will be administered orally, daily and continuously.
  Interventions: Drug: Bicalutamide

INTERVENTIONS:
Drug: Vandetanib — Vandetanib at 300 mg in combination with Bicalutamide at 50 mg will be administered orally, daily and continuously
  Arms: A
Drug: Bicalutamide — Bicalutamide at 50 mg will be administered orally, daily and continuously.
  Arms: B

SUMMARY:
Purpose To define the efficacy, tolerability and safety of Vandetanib in combination with bicalutamide in patients with chemotherapy naive hormone refractory prostate cancer

Hypothesis There will be a PSA response when Vandetanib is given in combination with Bicalutamide in Chemotherapy Naive Hormone refractory prostate cancer patients.

DETAILED DESCRIPTION:
With the advent of PSA surveillance, many patients diagnosed with hormone refractory disease, have PSA rising disease only, are asymptomatic, with no evidence of metastatic disease. There is no standard of care in this patient population. A standard treatment in this population has been the addition of a non-steroidal anti androgen such as bicalutamide. PSA response rate (defined as a 50% decrease) have been reported in 20% range with bicalutamide.

Even in patients with hormone refractory prostate cancer (HRPC) and metastases that have no cancer related symptoms, initiation of chemotherapy is controversial given the palliative nature of chemotherapy and potential for serious toxicity.

These patients are generally well enough to to undergo trials of novel agents and achieve adequate drug exposure, such that any cytostatic effect will be apparent.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a pathological diagnosis of adenocarcinoma of the prostate
* Patients must have biochemically recurrent disease or metastatic disease that is asymptomatic or minimally symptomatic (total daily morphine dose < 30mg.day) for which no curative therapy exists.
* Patients must have documented evidence od PSA progression while receiving androgen ablative therapy (i.e. must be hormone refractory). Progression is defined as the development of new metastatic lesions, or rising PSA defined as at least two rises in PSA at least 1 week apart. If the second PSA is not rising, a thrid PSA is required to show further increase; if not, a subsequent level must show further increase. The third (or subsequent) PSA confirming progression must be within 2 weeks of randomization.
* The PSA must be => 2ug/L at the time of study entry.
* ECOG performance status of 0 or 1
* Age =>18 years
* Patients must have a life expectancy of at least 12 weeks
* No Prior chemotherapy is permissible for hormone refractory disease. Chemotherapy may have been received in a neoadjuvant or adjuvant setting provided it was given 12 months prior to registration.
* Hormone Therapy

  * Prior hormone therapy in the form of either medical or surgical castration is required. If the patient is receiving medical androgen abalation a castrate level of testosterone (1.7nmol/L) must be present. Therapy with LHRH agonist must continue for those prostate cancer patients already receiving this treatment at the time of registration. If the patients has discontinued the LHRH agonist, this must be restarted and a castrate level of testosterone must be present.
  * Prior use of nonsteroidal antiandrogens (including bicalutamide) is permitted but must have been discontinued 6 weeks prior to registration.
* Prior external beam radiation is permitted provided a minimum of 4 weeks has elapsed between the last dose and registration in the trial. Exceptions will be made for limited field, single fraction palliative radiation to bone.
* No concurrent treatment with steriods unless steriods have been ingested for 4 weeks prior to commencing study at a dose of less than or equal to an equivalent of prednisone 20mg per day.
* No concurrent experimental trial medication is permitted. No prior use of VEGF/VEGFR or EGFR targeting agents for hormone refractory disease is permitted.
* Laboratory Requirements- within 7 calendar days prior to registration Hematology: haemoglobin >= 100g/L neutrophils >=1.5 x 10(9)/L Platelets >=100 x 10(9)/L INR =<1.5 x upper limit of normal Biochemistry: AST, ALT = <1.5 x upperlimit of normal Bilirubin <1.5 x upper limit of normal Serum creatinine <1.5 x upper limit of normal
* Baseline QTc (Bazett's) <480msec determined by the average of a least 3 consecutive electrocardiograms (ECG) taken within 5-10 mins of each other.
* Patient consent must be obtained according to local institutional and/or University Research and Ethic Board (REB) requirements.
* Patients must be accessible for treatment and follow up.
* Protocol treatment is to begin within 7 calendar days of patient registration.

Exclusion Criteria:

* Patients with a history of other invasive malignancy, except:adequately treated non melanoma skin cancer or other solid tumors curatively treated with no evidence of disease for 3 years.
* Patients with known brain metastases or leptomemingeal disease are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurological dysfunction that would confound the evaluation of nerologic and other adverse events.
* History of allergic reactions and/or sensitivity attributed to compounds of similar chemical or biological composition to Vandetanib or other agents used in the study.
* Other serious intercurrent illness or medical condition that might be aggravated by protocol treatment including;myocardial infarction within 6 months prior to study entry, congestive heart failure, unstable angina,cardiomyopathy, unstable ventricular arrhythmias,OTc (Bazett's) >480msec Uncontrolled hypertension (systolic >160, diatolic >100) Uncontrolled psychotic disorders, serious infections,peptic ulcer disease,history of bleeding diathesis
* Upper gasrtointerstinal or other conditions that would preclude compliance with oral medication
* Patients with immune deficiency are at increased risk of lethal infections when treated with Marrow-suppressive therapy. Therefore, HIV positive patients receiving combination ant-retroviral therapy are excluded from study because of possible risk of lethal infection and additionally because of the possible pharmacokinetic interactions with Vandetanib. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated.
* Patients who require escalating amounts of narcotic therapy to control pain e.g. morphine equivalent dose >30mg/day) since these patients would more appropriately be offered systemic chemotherapy
* Patients who require therapeutic anticoagulation with warfarin.
* Patients who require the following medication:concomittant use of warfarin, Class 1A antiarrythmics (e.g., quinidine, procainamide, disopyramide) Class

  1C antiarrhythmics (e.g.,flecainide, propafenone), Class III antiarrhythmics (e.g., amiodarone, sotalol, ibutilide), antipsychotics (e.g., thioridazine, chlorpromazine, pimozide, haloperidol, droperidol), tri/tetracyclic antidepressants (e.g., amitriptyline, imipramine, maprotiline), ketoconazole, antiepileptics and macrolide antibiotics.
* Patients who cannot stop ingestion of grapefruit/juice.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-01; Primary Completion 2012-02 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
PSA response | Continuous to end of study

SECONDARY OUTCOMES:
time to over all progression | continuous
Evaluation of treatment related toxicity | continuous

CONTACTS AND LOCATIONS:
Overall Officials: Kim Chi, MD, Study Chair — BC Cancer Agency - Vancouver Centre
Locations (4):
- Canada (4):
  - BC Cancer Agency - Centre for Southern Interior, Kelowna, British Columbia
  - BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario